CLINICAL TRIAL: NCT01035333
Title: A Pilot Study of the Efficacy of Alli in the Management of Pre-operative Weight Loss Required for Bariatric Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albany College of Pharmacy and Health Sciences (Other)
Collaborators: Albany Medical College (Other)
Responsible Party: Principal Investigator, Margaret Malone, Dr, Albany College of Pharmacy and Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-016
Record Dates: First submitted 2009-12-15; First posted 2009-12-18 (Estimated); Results first posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-02

CONDITIONS: Obesity
Keywords: gastric bypass surgery
MeSH Terms: conditions — Obesity | interventions — Orlistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- orlistat 60mg (Experimental): Patients assigned to treatment group for up to 6 months of therapy.
  Interventions: Drug: Orlistat

INTERVENTIONS:
Drug: Orlistat — 60mg capsule three times a day for up to 6 months
  Other Names: Alli

SUMMARY:
The primary goal of the study is to determine if orlistat 60mg (Alli) is effective in helping patients achieve a required 10% weight loss goal prior to bariatric surgery. The medication will be added to the usual standard of care which includes education regarding diet and exercise and monthly meetings with a registered dietician.

ELIGIBILITY:
Inclusion Criteria:

* adult patients preparing for gastric bypass surgery

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Malone, PhD, Principal Investigator — Albany College of Pharmacy and Health Sciences
Locations (1):
- Albany College of Pharmacy and Health Sciences, Albany, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment 10.14.09 to 12.15.10 Outpatient clinic, Bariatric treatment Center
Period: Overall Study
Arm/Group | Orlistat 60mg
Started | 19
Completed | 9
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Orlistat 60mg
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss
Description: Weight loss acheived during time on study up to 6 months.
Time Frame: 6 months
Population: All patients data who were entered were analyzed, 19 recruited, 15 at 3 months, 9 at 6 months.
Measure: Mean (Standard Deviation); unit: percentage of weight
Arm/Group | Orlistat 60mg
Number analyzed (Participants) | 9
percentage of weight | 2.0 (3.4)

2. Secondary Outcome: Patient Satisfaction
Time Frame: 6 months
Population: Patients who completed 6 months of the study.
Measure: Number; unit: participants
Arm/Group | Orlistat 60mg
Number analyzed (Participants) | 9
participants | 9

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Orlistat 60mg
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

LIMITATIONS AND CAVEATS:
High drop out rate. Patients did not return to clinic and were lost to follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No